CLINICAL TRIAL: NCT04956042
Title: A Phase 1B/2A, Open-label Study of the Safety, Pharmacokinetics, and Pharmacodynamics of Fosciclopirox Alone and In Combination With Cytarabine in Patients With Relapsed/Refractory Acute Myeloid Leukemia (AML)
Brief Title: Study of Fosciclopirox in Patients With Relapsed/Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Discontinued
Sponsor: CicloMed LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CPX-POM-003
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Refractory Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 - Fosciclopirox only (Experimental): An initial 14 study participants will be enrolled in Cohort 1a and will be treated with fosciclopirox. If there is a disease response, an additional 14 study participants will be enrolled into Cohort 1 (Cohort 1b).
  Interventions: Drug: Fosciclopirox
- Cohort 2 - Fosciclopirox + Cytarabine (Experimental): To be implemented if a disease response is not seen in Cohort 1a. Cohort 2a will have an initial 14 study participants treated with fosciclopirox and cytarabine. If a disease response is seen, an additional 14 study participants will be enrolled (Cohort 2b).
  Interventions: Drug: Fosciclopirox + Cytarabine

INTERVENTIONS:
Drug: Fosciclopirox — Fosciclopirox, 900 mg/m2 administered as a 20-minute IV infusion once daily on D1-D5 of each 21-day treatment cycle
  Arms: Cohort 1 - Fosciclopirox only
Drug: Fosciclopirox + Cytarabine — Fosciclopirox - 900 mg/m2 administered as a 20-minute IV infusion once daily on D1-D5 of each 21-day treatment cycle
  Cytarabine - 1g/m2 once daily on D1-D5 of each 21-day treatment cycle
  Arms: Cohort 2 - Fosciclopirox + Cytarabine

SUMMARY:
This will be an open-label, Phase 1B/2A, study to characterize the efficacy, safety, pharmacokinetics, and pharmacodynamics of fosciclopirox administered alone and in combination with cytarabine in patients with R/R AML with up to two cohorts studied to confirm the efficacy (or futility) of fosciclopirox on the endpoint of disease response.

Initially, 14 evaluable patients will be enrolled in Cohort 1a. If disease response to fosciclopirox alone IS observed in at least 4 of 14 patients, an additional 14 patients will be enrolled in Cohort 1b. If disease response to fosciclopirox alone IS NOT observed in at least 4 of 14 patients in Cohort 1a, based on a review of all available study data, the study may be terminated OR a Cohort 2a may be initiated using the combination of fosciclopirox and cytarabine. If disease response to fosciclopirox in combination with cytarabine IS observed in at least 4 of 14 patients in Cohort 2a, an additional 14 patients will be enrolled in Cohort 2b. If disease response to fosciclopirox in combination with cytarabine IS NOT observed in at least 4 of 14 patients in the Cohort 2a, the study will be stopped for futility.

DETAILED DESCRIPTION:
This will be an open-label, Phase 1B/2A, study to characterize the efficacy, safety, PK, and pharmacodynamics of fosciclopirox administered alone and in combination with cytarabine in patients with R/R AML. There will be up to two cohorts used to confirm the efficacy (or futility) of fosciclopirox on the endpoint of disease response.

Initially, 14 patients will be enrolled in Cohort 1a. If disease response to fosciclopirox alone IS observed in at least 4 of 14 patients, an additional 14 patients will be enrolled in Cohort 1b. If disease response to fosciclopirox alone IS NOT observed in at least 4 of 14 patients in the initial Cohort 1a, based on a review of all available data study data, the study may be terminated OR a second cohort (Cohort 2a) may be initiated using the combination of fosciclopirox and cytarabine. If disease response to fosciclopirox in combination with cytarabine IS observed in at least 4 of 14 patients in Cohort 2a, an additional 14 patients will be enrolled in Cohort 2b. If disease response to fosciclopirox in combination with cytarabine IS NOT observed in at least 4 of 14 patients in Cohort 2a, the study will be stopped for futility.

If both Cohorts 1a and 2a are initiated, the minimum patient number will be 28 (i.e., treatment with fosciclopirox alone and in combination with cytarabine are futile). The maximum number of patients potentially evaluated is 42 (i.e., the first treatment is futile based upon observations in 14 patients (Cohort 1a), but treatment in Cohort 2a evaluated is positive [14 patients], and Cohort 2b [14 patients] is completed).

Patients in Cohort 1a will initially be treated with fosciclopirox as a single agent. Patients who respond to this treatment, as defined below, may continue to receive treatment cycles of fosciclopirox alone until evidence of disease progression. Patients who do not respond to fosciclopirox alone, as defined below, may be switched to treatment with the combination of fosciclopirox and cytarabine. Patients who respond to the combination treatment may continue to receive treatment cycles of fosciclopirox in combination with cytarabine until evidence of disease progression. Patients who do not respond to the combination of fosciclopirox and cytarabine will be discontinued from the study.

Patients enrolled in Cohort 2a (if initiated) will initially be treated with fosciclopirox in combination with cytarabine. The first patient to receive this combination will be observed during Cycle 1 (21 days) and for a further 7 days (if they do not continue to Cycle 2) before any further patients are accrued to the combination arm. As above, patients who respond to the combination treatment may continue to receive treatment cycles until evidence of disease progression, and patients who do not respond will be discontinued from the study.

Fosciclopirox will be administered as 900 mg/m2 once daily as a 20-minute intravenous infusion on Days 1 to 5 (D1-D5) of each 21-day treatment cycle (rest days D6-D21). When added to fosciclopirox therapy, cytarabine will be administered as 1 gm/m2 once daily on D1 D5 of each 21-day treatment cycle (rest days D6-D21).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female aged ≥18 years.
2. Patient provided signed and dated informed consent prior to initiation of any study procedures.
3. Patient has relapsed AML after complete remission of any duration as evidenced by presence of neoplastic blasts in the bone marrow confirmed by flow cytometry OR has refractory AML, defined as primary refractory to at least 2 cycles of induction therapy.
4. No other therapy exists or patient has received all standard therapies that would be potentially curative or might provide significant benefit.
5. Patient has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0, 1, or 2.
6. Patient has a predicted life expectancy of ≥3 months.
7. Patient has a total white blood cell count of count ≤ 25.0 x 10^9/L at screening and on C1D1. (Patient may have received hydroxyurea prior to the screening sample for elevated WBC but must have discontinued the therapy at least 72 hours prior to screening, and not be treated with hydroxyurea after the screening sample has been taken).
8. Patient has adequate renal function (creatinine ≤2 × the upper limit of the normal range (ULN) and an estimated glomerular filtration rate (eGFR) of >30 mL/min/1.73 m^2).
9. Patient has adequate hepatic function, as evidenced by a total bilirubin ≤2 × ULN, aspartate aminotransferase (AST) ≤5 × ULN and /or alanine aminotransferase (ALT)

   ≤5 × ULN, unless due to leukemia involvement in the judgement of the Principal Investigator in consultation with the Medical Monitor.
10. Patient has adequate cardiac function with an ejection fraction (EF) ≥45%, as assessed by multi-gated acquisition (MUGA) or ultrasound/echocardiography (ECHO) and corrected QT interval by Fridericia's correction formula (QTcF) <450 msec for males and <470 msec for females. The eligibility of patients with ventricular pacemakers for whom the QT interval may not be accurately measurable will be determined on a case-by-case basis by the Sponsor in consultation with the Medical Monitor.
11. Patient and his/her partner agree to use adequate contraception after providing written informed consent through 3 months after the last dose of fosciclopirox, as follows:

    1. For women: Negative pregnancy test during Screening and at Day 1 of each treatment cycle and compliant with a medically-approved contraceptive regimen during, and for 3 months after, the Treatment period or documented to be surgically sterile or postmenopausal.
    2. For men: Compliant with a medically-approved contraceptive regimen during, and for 3 months after, the Treatment period or documented to be surgically sterile. Men whose sexual partners are of child-bearing potential must agree to use 2 methods of contraception prior to study entry, during the study, and for 3 months after the Treatment period. Men must also agree not to donate sperm during the Treatment period and for 3 months after the Treatment period.
12. Patient is willing and able to participate in the study and comply with all study requirements.
13. Prior allogeneic stem cell transplant is allowed as long as patient is more than 100 days post-transplant and has no active graft versus host disease.

Exclusion Criteria:

Patients who meet any of the following exclusion criteria are not to be enrolled in this study.

1. Patient has another active malignancy.
2. Patient has acute promyelocytic leukemia (APL) or Ph+ AML.
3. Patient has total white blood cell count >25.0 x 10^9/L at C1D1.
4. Patient has clinically significant cardiac disease.
5. Patient has known chronic active liver disease or evidence of acute or chronic Hepatitis B Virus (HBV) or Hepatitis C (HCV).
6. Patient has known diagnosis of human immunodeficiency virus (HIV) infection. Testing is not required in absence of clinical suspicion.
7. Patients has any serious and/or uncontrolled concurrent medical conditions (e.g., uncontrolled infection, uncontrolled diabetes) or psychiatric illness that could, in the investigator's opinion, cause unacceptable safety risks or potentially interfere with the completion of the treatment according to the protocol.
8. Patient has received any live viral vaccine used for prevention of infectious diseases within 4 weeks prior to Baseline.
9. If female, patient is pregnant or breast-feeding.
10. Patient is taking warfarin.
11. Patient has known allergy or hypersensitivity to any component of fosciclopirox.
12. Patient is taking any iron replacement therapy administered IV, intramuscularly, or orally due to the potential for loss of anticancer activity due to drug and/or metabolites chelating iron.
13. Patient is taking Hydrea (hydroxyurea) within 72 hours prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Acute Myeloid Leukemia (AML) response | Screening through Day 42
  Complete remission [CR], CR with incomplete hematologic recovery [CRi], partial remission [PR], or morphologic leukemia-free state [MLFS] at the conclusion of the first treatment cycle OR Nonprogression at the end of the first treatment cycle (defined as no increase in bone marrow or peripheral blood blast count) followed by CR, CRi, PR, or MLFS at the conclusion of the second treatment cycle
Frequency and type of treatment-related AEs | From Informed Consent Form through Follow Up visit (30±5 days after last dose of study drug)
  Adverse events as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - John Hopkins School of Medicine, Baltimore, Maryland